CLINICAL TRIAL: NCT00460096
Title: Randomized Double-Blind Comparison of an Alpha-1 Proteinase Inhibitor (Kamada API) With a Currently Marketed API Product in Individuals With Alpha-1 Antitrypsin Deficiency
Brief Title: Phase II/III Study of an Alpha-1 Proteinase Inhibitor (Kamada-API) in Individuals With Alpha-1 Antitrypsin Deficiency
Acronym: Kamada API
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Kamada, Ltd. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Kamada API-002
Record Dates: First submitted 2007-04-12; First posted 2007-04-13 (Estimated); Last update posted 2007-10-17 (Estimated); Status verified 2007-10

CONDITIONS: Alpha 1-Antitrypsin Deficiency
Keywords: Pulmonary Emphysema
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Pulmonary Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Kamada-API

SUMMARY:
The primary purpose of this Phase II/III study is to demonstrate that Kamada-API, a new API concentrate manufactured by Kamada Ltd., is comparable to a currently marketed API product.

DETAILED DESCRIPTION:
Alpha-1 Antitrypsin Deficiency, also called Alpha-1-Proteinase Inhibitor (API) deficiency, is a genetic disorder characterized by the production of an abnormal amount of AAT protein and reduced circulating levels of this protein. Subjects with AAT deficiency are at increased risk for developing chronic obstructive pulmonary disease (COPD). It is believed that this is the result of the chronic activity of elastase released by cells continually present in the lungs in low numbers.

This study is a randomized, double-blind comparison of Kamada API, an Alpha-1-Proteinase Inhibitor with a currently marketed API product.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. "At-risk" alleles associated with serum AAT < 11 μM including null alleles and deficiency alleles. This must be documented in the subject's history or laboratory tests performed at screening.
3. At least 18 years of age.
4. Evidence of lung disease related to AAT deficiency, identified by at least one of the following:

   * FEV1<80% predicted (post BD); or
   * Loss of lung function over a one year period of greater than 35ml in FEV1; or
   * HRCT evidence of pulmonary emphysema
5. For actively treated subjects, agreement to not receive any exogenous API product (i.e. washout) for five weeks prior to first study infusion.
6. Use of an effective means of contraception during the 24 weeks of study drug administration (this is applicable to both sexes).
7. Subjects on the BAL, bronchial brushing/biopsy group must be on inhaled corticosteroids at a stable dose two weeks prior the first Bronchoscopy and throughout the dosing period up the final bronchoscopy.

Exclusion Criteria:

1. Laboratory evidence of severe IgA deficiency (from medical history or by IgA testing at screening of at least 20% of lower range).
2. Current smoker or a history of smoking within the past 3 months.
3. History of allergy to plasma proteins.
4. Participation in another experimental drug or device trial within the past 30 days.
5. Evidence of uncontrolled hypertension (systolic ≥180 mm Hg, and/or diastolic ≥ 110 mm Hg on 3 consecutive occasions in the supine position)
6. Pulse ≥ 120/min (prior to the 1st infusion).
7. Abnormal screening or baseline laboratory measurements that in the opinion of the Investigator would affect subject safety.
8. Pregnancy or lactation.
9. Current life-threatening malignancy.
10. Previous organ transplant recipient.
11. History of infection with HCV, HBV and/or HIV 1 or 2, or (at baseline) infection indicated by laboratory measurements obtained at screening.
12. Acute respiratory tract infection or COPD exacerbation which required antibiotic and/or systemic steroid treatment within the past 6 weeks. Patient can be re-evaluated for enrollment 6 weeks after an exacerbation.
13. Any other condition which in the judgment of the investigator may interfere with the conduct of the study.
14. If an adequate home health care agency cannot be established by Centric Health Resources due to a potential subject's geographical location.

Exclusion criteria for subjects entering into the BAL and bronchial biopsy/brushing:

1. FEV1 < 45% predicted (post-BD).
2. Inability to undergo bronchoscopy.
3. Allergy to lidocaine.
4. Exacerbation of COPD in the previous 6 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-03; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Efficacy

SECONDARY OUTCOMES:
Safety

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Sandhaus, M.D., Principal Investigator — National Jewish Health
Locations (3):
- United States (3):
  - National Jewish Medical and Research Center, Denver, Colorado
  - University of Florida School of Medicine, Gainesville, Florida
  - The University of Texas Health Center at Tyler, Tyler, Texas

REFERENCES:
- [Derived] Sandhaus RA, Stocks J, Rouhani FN, Brantly M, Strauss P. Biochemical efficacy and safety of a new, ready-to-use, liquid alpha-1-proteinase inhibitor, GLASSIA (alpha1-proteinase inhibitor (human), intravenous). COPD. 2014 Feb;11(1):17-25. doi: 10.3109/15412555.2013.804500. Epub 2013 Jul 3. PMID 23822603